CLINICAL TRIAL: NCT02387099
Title: A Multicenter, Randomized, Double-blind, Phase II Study to Evaluate the Tolerability of an Induction Dose Escalation of Everolimus in Patients With Metastatic Breast Cancer
Brief Title: Dose EScalation Induction of EvERolimus
Acronym: Desiree
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBG 86
Record Dates: First submitted 2015-03-05; First posted 2015-03-12 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer; Hormone Receptor Positive Tumor
Keywords: Stage IIIB; Stage IV; Recurrent; Metastatic
MeSH Terms: conditions — Breast Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Everolimus dosing according to label (Active Comparator): everolimus 10 mg/day, week 1-3: 4x2.5 mg/day (blinded); week 4-24: 10mg/day (open according to label)
  + further treatment according to standard of care
  Interventions: Drug: 3 weeks Conventional Everolimus Dosing; Drug: Open Label Phase with conventional 10mg Everolimus Dosing week 4-24; Drug: Standard Care after 24 weeks
- 3 week Dose Induction of Everolimus (Experimental): an escalating dose of everolimus as follows: week 1: 1x2.5 mg verum + 3x placebo/day; week 2: 2x2.5 mg verum + 2x placebo/day; week 3: 3x2,5 mg verum + 1x placebo/day; week 4-24: 10 mg/day (open according to label)
  + further treatment according to standard of care
  Interventions: Drug: 3 weeks Dose Induction of Everolimus; Drug: Open Label Phase with conventional 10mg Everolimus Dosing week 4-24; Drug: Standard Care after 24 weeks

INTERVENTIONS:
Drug: 3 weeks Dose Induction of Everolimus — Comparing a conventional dosing approach starting with 10 mg at first dose versus a dose-escalating schema over 21 days in patients receiving everolimus in combination with exemestane for treatment of metastatic breast cancer.
  All patients will be treated within the approved indication of everolimus in combination with exemestane.
  Patients will be randomized in a 1:1 ratio
  Arms: 3 week Dose Induction of Everolimus
Drug: 3 weeks Conventional Everolimus Dosing — Comparing a conventional dosing approach starting with 10 mg at first dose versus a dose-escalating schema over 21 days in patients receiving everolimus in combination with exemestane for treatment of metastatic breast cancer.
  All patients will be treated within the approved indication of everolimus in combination with exemestane.
  Patients will be randomized in a 1:1 ratio
  Arms: Conventional Everolimus dosing according to label
Drug: Open Label Phase with conventional 10mg Everolimus Dosing week 4-24 — All patients will receive open label Everolimus with Exemestane for 21 weeks according to label
Drug: Standard Care after 24 weeks — It is up to the discretion of the investigator to continue with Everolimus+Exemestane beyond 24 weeks

SUMMARY:
The BOLERO-2 study demonstrated a benefit for patients who received everolimus in addition to exemestane in patients who progressed during/after a non-steroidal aromatase inhibitor;

Routine use of everolimus shows an high rate of intolerability due to mucositis/stomatitis especially during the first 12 weeks of treatment leading cause for treatment discontinuation not related to tumor progression;

GeparQuinto study (setting III: non-responders): everolimus was given as salvage treatment in combination with paclitaxel for patients without response to 4 cycles epirubicin/cyclophosphamide with/without bevacizumab.

A dose-escalation schema was successfully used to improve tolerability of everolimus together with the cytotoxic Agent.

Everolimus plus exemestane has improved the prognosis of metastatic breast cancer significantly. Desiree-study aims to improve the tolerability, which is necessary in order to achieve an adequate dose intensity for the patients in Routine care.

DETAILED DESCRIPTION:
The BOLERO-2 study demonstrated an enormous benefit for patients who received everolimus in addition to exemestane in patients who progressed during/after a non steroidal (NSAI), which led to approval of everolimus in this indication. However, experience from routine use report a high rate of intolerability of this innovative treatment approach especially during the first 12 weeks of treatment. Most common side effect is mucositis/Mucositis which is considered the leading cause for treatment discontinuation not related to tumor progression.

This outside clinical trial experience is contrary to findings from BOLERO-2, where the number of patients still taking full-dose (10mg) of everolimus at 4, 8, and 12 weeks is 77.8%, 75.6%, and 75.6%, respectively. These findings are in concordance with non-interventional studies. However, findings might be biased by positive pre-selection.

In the non-responder part (setting III) of the neoadjuvant GeparQuinto study, everolimus was given as salvage treatment in combination with paclitaxel for patients without response to 4 cycles epirubicin/cyclophosphamide +/- bevacizumab. A dose-escalation schema was successfully used to improve tolerability of everolimus together with the cytotoxic agent. In fact the addition of everolimus to paclitaxel led only to increases of grades 1-4 leukopenia, grades 1-2 thrombocytopenia, leukopenia, skin changes and hyperlipidemia. Grades 3-4 hematological and nonhematological toxic effects were infrequent with no differences between treatment arms.

Moreover, Ravaud et al performed a metaanalysis of clinical trials in order to evaluate the potential relationship between everolimus exposure, safety and efficacy. Previous studies have shown that maximum everolimus concentrations are reached 1-2 hours after administering 5-70 mg oral doses, maximum everolimus concentrations increase in a dose-proportional manner between 5 mg and 10 mg and that continuous 5-10 mg once-daily dosing enables steady state to be achieved within 1 week.

The metaanalysis shows that a two-fold increase in the minimum concentration of everolimus increased the probability of tumor size reduction (odds ratio 1.4), which was associated with a trend for reduced risk of PFS events (risk ratio [RR] 0.9), but with an increased risk of grade 3 pulmonary toxicity (RR1.93), Mucositis (RR 1.49), and metabolic toxicity (RR 1.3).

Taking together these results suggest a dose-dependent antitumor effect of everolimus that have to be balanced against the correlated increased toxicities. For this reason the optimal dose and schedule need to be explored within randomized prospective clinical trial, in order to increase compliance and tolerability, maximizing efficacy.

ELIGIBILITY:
Eligibiltiy according to Everolimus label (ie. postmenopausal women)

Inclusion Criteria (most important)

* Locally advanced or metastatic stage of disease not amenable to curative treatment by surgery or radiotherapy alone.
* No indication for chemotherapy (e.g. symptomatic visceral metastasis) -Histological confirmed hormone receptor-positive (HR+), HER2- negative carcinoma of the breast.
* Postmenopausal women
* Disease progression following prior therapy with non steroidal aromatase inhibitors (NSAI), defined as:

  1. Recurrence while on, or following completion of an adjuvant treatment with Letrozole or Anastrozole, or
  2. Progression while on or following completion of Letrozole or Anastrozole treatment for ABC/MBC. Note: Non-steroidal aromatase inhibitors (i.e. Letrozole or Anastrozole) do not have to be the last treatment prior to enrollment. Other prior anticancer therapy, e.g. Tamoxifen, Fulvestrant, Exemestane, is also allowed. Patients must have recovered to grade 1 or better from any adverse events (except alopecia) related to previous therapy prior to enrollment.
* At least 4 weeks since radiotherapy, with full recovery. The measurable disease must be completely outside the radiation field or there must be pathologic proof of newly progressive disease.

Exclusion Criteria (most important):

* Concurrent immunotherapy or hormonal therapy (contraceptive and/or replacement therapy). Bisphosphonates or denosumab may be continued or started before randomization.
* Life expectancy of less than 3 months.
* Parenchymal brain metastases, unless adequately controlled by surgery and/or radiotherapy.
* Any ongoing toxicity from prior anti-cancer therapy that is grade 3-4 and/or that is progressing in severity, except alopecia or anemia controlled by growth factors.
* Known or suspected congestive heart failure (>NYHA I) and/or coronary heart disease, angina pectoris requiring anti-anginal medication, previous history of myocardial infarction ≤ 6months, evidence of transmural infarction on ECG, un- or poorly controlled arterial hypertension (i.e. BP >150/100 mmHg under treatment with two antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease.
* Currently active infection.
* History of other malignancies within the last 5 years which significantly affect the diagnosis, assessment or prognosis of metastatic breast cancer.
* Malabsorption syndrome or insufficient gastrointestinal function, preexisting diagnosis of ulcerative colitis.
* Concurrent treatment with other experimental drugs; participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
* Insufficiently controlled diabetes, known HIV infection or chronic hepatitis B or C and seriously impaired liver function (Child-Pugh, class A, B or C).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-05; Primary Completion 2021-05 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
cumulative rate Mucositis grade 2-4 (WHO's oral toxicity scale (OTS)) | week1 to week 12
  To compare the cumulative rate of mucositis/stomatitis grade 2-4 (WHO's oral toxicity scale (OTS)) at 12 weeks after start of treatment using a conventional and a dose-escalating schema of everolimus in combination with exemestane in patients with metastatic breast cancer and progression or relapse after non-steroidal aromatase-inhibitor treatment.
  Endpoint measurement: First episode of mucositis WHO's OTS 2-4 any time during a 12 week period after start of everolimus

SECONDARY OUTCOMES:
cumulative rate Mucositis grade 2-4 (WHO's oral toxicity scale (OTS)) | week 1 to 24
  To compare the cumulative rate of mucositis/stomatitis grade 2-4 (WHO's oral toxicity scale (OTS)) at 24 weeks after start of treatment.
  Incidence of first episodes of mucositis/stomatitis WHO's OTS grade 2-4 any time during a 24 week period.
cumulative rate Mucositis any grade (WHO's oral toxicity scale (OTS)) | week 1 to 12 and week 1 to 24
  To compare the cumulative rate of mucositis/stomatitis grade 1 and any grade (WHO's oral toxicity scale (OTS)) at 12 and 24 weeks after start of treatment.
  Incidence of first episodes of mucositis/stomatitis WHO's OTS grade 1 and any grade any time during a 12 and 24 week period.
Patients on conventional dose Everolimus 10mg | week 12 and week 24
  To compare the rate of patients on 10mg daily at 12 weeks and 24 weeks after start of everolimus treatment. Average dose of treatment during week 12 and during week 24.
Clinical Benefit Rate (CBR) | week 24
  To compare the clinical benefit rate (CR, PR und SD >=16 Weeks) at 24 weeks after start of everolimus treatment. Clinical benefit rate (CBR) is defined as all patients with no evidence for tumor progression at 24 weeks after start of everolimus treatment.
Safety other than Mucositis | week 1 to 24
  To compare the safety with regard to other organ signs and symptoms.Safety by toxicity grades in general is defined by the NCI-CTCAE version 4.03.
Time to Mucositis grade 2-4 (WHO's oral toxicity scale (OTS)) | week 1 to 24
  To compare the time to grade ≥2 mucositis/stomatitis
Cumulative Dose | week 4
  To compare the cumulative dose at 4 weeks
RDI | week 1 to 24
  To compare the relative dose intensity for everolimus. Relative dose intensity for everolimus is the ratio of Actual Total Dose Intensity (ATDI) and Planned Total Dose Intensity (PTDI), expressed as a percentage.
QoL FACTB | week 4, week 12, End of Therapy Visit (week 25-28)
  To compare quality of life using the FACT-B questionnaire and the QSDQ
QoL QSDQ | daily till week12
  To compare quality of life using the FACT-B questionnaire and the QSDQ

OTHER OUTCOMES:
Biomarker for Breast Cancer | Baseline and End of Therapy Visit (week 25-28)
  Other objectives:
  Potential biomarkers predicting safety and compliance will be determined after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Loibl, Prof., MD, Study Chair — ASCO, ESGO, ESMO, DKG, DGGG, AGO, DGS, BIG, BCIRG, St. Gallen Faculty Member, SABCS Faculty member
Locations (14):
- Germany (14):
  - Sana Klinikum Offenbach / German Breast Group, Neu-Isenburg, Hesse
  - TU Dresden, Dresden, Saxony
  - Bielefeld
  - Cologne
  - University of Erlangen, Erlangen
  - Essen
  - Goslar
  - Hanau
  - Karlsruhe
  - Kiel
  - Mainz
  - München
  - Rotenburg (Wümme)
  - Weinheim

REFERENCES:
- [Derived] Schmidt M, Lubbe K, Decker T, Thill M, Bauer L, Muller V, Link T, Furlanetto J, Reinisch M, Mundhenke C, Hoffmann O, Zahn MO, Muller L, Denkert C, van Mackelenbergh M, Fasching PA, Burchardi N, Nekljudova V, Loibl S. A multicentre, randomised, double-blind, phase II study to evaluate the tolerability of an induction dose escalation of everolimus in patients with metastatic breast cancer (DESIREE). ESMO Open. 2022 Dec;7(6):100601. doi: 10.1016/j.esmoop.2022.100601. Epub 2022 Nov 7. PMID 36356410
- See also: Desiree website on German Breast Group home portal — https://www.gbg.de/de/studien/desiree.php